CLINICAL TRIAL: NCT02455921
Title: Comparative Effect of Neuromuscular Blockade Reversal Agent on Extubation Conditions, Postoperative Cognitive Function and Behaviour of School-aged Children Undergoing Ear Note Throat (ENT) Surgery
Brief Title: Neuromuscular Blockade Reversal Agent Effect on Postoperative Cognitive Function and Behaviour in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Associate Professor of Anaesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: EBD 712/19-3-15
Record Dates: First submitted 2015-05-20; First posted 2015-05-28 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Anesthesia; Functional
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sugammadex (Active Comparator): iv sugammadex 2 mg/Kg
  Interventions: Drug: Sugammadex
- neostigmine - atropine (Active Comparator): iv neostigmine 0,05 mg/Kg - atropine 0,02 mg/kg
  Efficacy, safety and effect on cognitive and behavioural function
  Interventions: Drug: neostigmine - atropine

INTERVENTIONS:
Drug: neostigmine - atropine — Efficacy, safety and effect on cognitive and behavioural function
  Arms: neostigmine - atropine
Drug: Sugammadex — Efficacy, safety and effect on cognitive and behavioural function
  Other Names: Bridion
  Arms: sugammadex

SUMMARY:
The aim of this prospective randomized study is to investigate comparatively the effect of neostigmine-atropine versus sugammadex on speed and quality of recovery and on postoperative cognitive function & behavior in children undergoing ENT surgery under general anaesthesia.

DETAILED DESCRIPTION:
The aim of this prospective randomized study is to investigate comparatively the effect of neostigmine-atropine vs sugammadex on time of achieving extubation, quality of recovery, postoperative cognitive function and behaviour of children undergoing ENT surgery under general anaesthesia.

In this study after parental approval has been obtained, children with age 6-12 yrs undergoing tonsillectomy and/or adenoidectomy under general anaesthesia will be included. General anaesthesia will be performed using Total Intravenous Anaesthesia (TIVA) technique with continuous infusion of propofol and remifentanil. Rocuronium will be used to achieve neuromuscular blockade (NMB). Neuromuscular reversal will be performed using either atropine-neostigmine or sugammadex. Patients will be divided into 2 groups according to the type of NMB reversal agent used. Intraoperative monitoring will include Bispectral Index Sedation (BIS), SpO2, capnography, noninvasive measurements of blood pressure, heart rate and train of four (TOF).

Children will be assessed preoperatively (one day before surgery and at the morning of day of surgery), intraoperatively, immediate postoperatively and will be followed up for 15 postoperative days. Additionally, parents will be cooperated and questioned.

The primary end-points of the study include the comparative investigation of the effect of neostigmine-atropine vs sugammadex on time of achieving extubation, quality of recovery, and postoperative cognitive function of children. Secondary endpoints will include side effects, signs of residual neuromuscular blockade, agitation and postoperative behavioural changes of children.

For this purpose the following scales and questionnaires will be used:

1. Emotionality, Activity, Sociability & Impulsivity (EASI) Scale
2. The Modified Mini-Mental State (3MS) Test - Version G Greek
3. Yale Preoperative Anxiety Scale
4. Aldrete score
5. Emergence Delirium (PAED) scale
6. Wong-Baker scale
7. Visual Analogue Scale (VAS) (0-10)
8. Child Post- Hospital Behavior Questionnaire (PHBQ)]
9. Post discharge repeated questionnaire

All the questionnaires will be translated, culturally adapted and validated in Greek. Analysis of the data will include pair wise T test in order to find statistical differences between the two techniques and regression analysis models in order to revile significant correlations between dependent and independent variables. Statistical analysis will be performed with the use of SPSS21 for Windows.

ELIGIBILITY:
Inclusion Criteria:

- Children undergoing ENT surgery under general anaesthesia.

Exclusion Criteria:

* Parents refusal
* Cognitive impairment
* Difficulty in communication due to language issues
* Psychiatric disorder
* Severe systematic disorder
* Known allergy to any drug used

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
time of achieving extubation | 10 min
  time of achieving extubation

SECONDARY OUTCOMES:
signs of residual neuromuscular blockade | 1 hour
  number of participants with signs of residual
Behavioural function | up to 15th postoperative day
  changes using Battery test

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi C Matsota, Assoc. Prof., Principal Investigator — 2nd Department of Anesthesiology, Attikon University Hospital Athens, Attiki Greece
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glinka L, Onichimowski D, Sieniuta P, Korecki A. [Sugammadex--two years in clinical practice]. Anestezjol Intens Ter. 2010 Jul-Sep;42(3):155-9. Polish. PMID 21413422